CLINICAL TRIAL: NCT04465422
Title: Development and Validation of the Client Centered Occupational Therapy Service Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCHIRB-10904021
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-06

CONDITIONS: Occupational Therapy; Psychiatric Rehabilitation
Keywords: client-centered; Model of Human Occupation
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: We will recruit 70 inpatients with schizophrenia and devided into intervention group, based on MOHO theory, and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blind during this clinical trial. They are prevented from having knowledge of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): We will recruit 70 inpatients with schizophrenia and divided into intervention group and control group. The Intervention group provided Occupational therapy based on the MOHO theory, while the control group adopted the original Occupational therapy model.
  The research at this stage is based on the theoretical framework of the MOHO model and the clinical practice of OTPF-3. Clinical experts are requested to assist in providing relevant suggestions as a reference for modifying intervention activities. Design OT@tcpc service model for occupational therapy intervention activities. The event design is based on the 4 systems of determinationl, habits, performance and environment, and 2 events are designed for each to be carried out in a group. Each activity includes 4 parts: warm-up, activity, feedback and homework. Each activity group will be explained separately so that the occupational therapist of the group can complete it under the guidance.
  Interventions: Behavioral: Occupational therapy based on the MOHO theory
- Control Group (Active Comparator): We will recruit 70 inpatients with schizophrenia and divided into intervention group and control group. The Intervention group provided Occupational therapy based on the MOHO theory, while the control group adopted the original Occupational therapy model.
  This study was approved by the Institutional Review Board of Taipei City Hospital. After informed consent, the patients signed the consent form for this study and became the participant of this study.
  Each activity group will be explained separately so that the participants of each group can complete it under the guidance. The group description includes: activity title, activity time (location), MOHO theory system, group purpose, activity content, equipment or materials, precautions, etc.
  Interventions: Behavioral: Occupational therapy

INTERVENTIONS:
Behavioral: Occupational therapy based on the MOHO theory — We selected two acute wards in the Songde hospital as the intervention group and the control group. At the same time, the demographic data of the participants were collected, including gender, age, age of onset, marital status, education level, work experience, etc., and the clinical records, including assessment of mental symptoms and medication records, etc. Continuity or categorical information on Occupational performance, personal and social performance, instrumental activities daily living, and clinical performance.
  OPHI-II, CGIS, PSP, LIADL, COPM, COTES were tested before and after in the intervention group and the control group to explain the intervention effect of the MOHO theory-based treatment model.
  Arms: Intervention Group
Behavioral: Occupational therapy — The original Occupational therapy. OPHI-II, CGIS, PSP, LIADL, COPM, COTES were tested before and after in the intervention group and the control group to explain the intervention effect of the MOHO theory-based treatment model.
  Arms: Control Group

SUMMARY:
The purpose of the study is to develop and validate Client-centered Occupational Therapy Service at Taipei City Psychiatric Center (OT@tcpc) service model to assist clinicians to provide and integrate comprehensive OT services.

DETAILED DESCRIPTION:
Occupational Therapy (OT) is one of the mental health services. The service phase includes acute/chronic hospitalization, daycare centers (adolescents, adults, and the elderly), community mental rehabilitation institutions, psychiatric nursing home, and outpatient assessment/treatments. OT provides holistic and continuous mental rehabilitation services at each stage of mental health care. During the acute hospitalization and based on the Model of Human Occupation (MOHO) model, the occupational therapist provides daily activities to assist acute patients with mental illness to develop occupation adaptation to enable and prepare for discharge.

However, the lack of a client-centered OT service model limits the interpretation of the treatment effect and the process of change. This will seriously affect the integrity and continuity of OT services and will limit the development of OT professions. Thus, the purpose of the study is to develop and validate Client-centered Occupational Therapy Service at Taipei City Psychiatric Center (OT@tcpc) service model to assist clinicians to provide and integrate comprehensive OT services.

This project consists of 2 stages. First, based on the MOHO model we use 5 stages with 6 weeks program to develop the OT@tcpc service model. Second, validate the to indicate the occupation identity and competence to validate the OT@tcpc service model. We will recruit 70 inpatients with schizophrenia and divided into intervention group, based on MOHO theory, and control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with schizophrenia according to DSM-5 diagnostic criteria.
2. Over 20 years old.
3. Agree to participate in the study

Exclusion Criteria:

* 1. Diagnosis of intellectual developmental disorders 2. History of severe brain injury 3. Cannot complete the study due to poor cognitive, vision or hand function

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Lee, Master, Principal Investigator — Department of Occupational Therapy
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee J. Achieving best practice: a review of evidence linked to occupation-focused practice models. Occup Ther Health Care. 2010 Jul;24(3):206-22. doi: 10.3109/07380577.2010.483270. PMID 23898928
- [Background] Lee SW, Taylor R, Kielhofner G, Fisher G. Theory use in practice: a national survey of therapists who use the Model of Human Occupation. Am J Occup Ther. 2008 Jan-Feb;62(1):106-17. doi: 10.5014/ajot.62.1.106. PMID 18254437
- [Background] Lee SW, Kielhofner G, Morley M, Heasman D, Garnham M, Willis S, Parkinson S, Forsyth K, Melton J, Taylor RR. Impact of using the Model of Human Occupation: a survey of occupational therapy mental health practitioners' perceptions. Scand J Occup Ther. 2012 Sep;19(5):450-6. doi: 10.3109/11038128.2011.645553. Epub 2012 Jan 3. PMID 22214401
- [Background] Melton J, Forsyth K, Metherall A, Robinson J, Hill J, Quick L. Program Redesign Based on the Model of Human Occupation: Inpatient Services for People Experiencing Acute Mental Illness in the UK. Occup Ther Health Care. 2008;22(2-3):37-50. doi: 10.1080/07380570801989382. PMID 23941371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of the recruitment period : 06/19/2020 - 07/16/2020 Recruitment type of location : medical clinical
Groups:
- Intervention Group: We will recruit 70 inpatients with schizophrenia and divided into intervention group and control group. The Intervention group provided Occupational therapy based on the MOHO theory.
  Occupational therapy based on the MOHO theory: We selected two acute wards in the Songde hospital as the intervention group and the control group. At the same time, the demographic data of the participants were collected, including gender, age, age of onset, marital status, education level, work experience, etc., and the clinical records, including assessment of mental symptoms and medication records, etc. Continuity or categorical information on Occupational performance, personal and social performance, instrumental activities daily living, and clinical performance.
- Control Group: We will recruit 70 inpatients with schizophrenia and divided into intervention group and control group. The control group adopted the original Occupational therapy model. Execution for two weeks.
  At the same time, the demographic data of the participants were collected, including gender, age, age of onset, marital status, education level, work experience, etc., and the clinical records, including assessment of mental symptoms and medication records, etc. Continuity or categorical information on Occupational performance, personal and social performance, instrumental activities daily living, and clinical performance.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 17 | 16
Completed | 17 | 14
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: In order to indicate the occupation identity and competence to validate the OT@tcpc service model. We recruited 70 inpatients with schizophrenia and divided into intervention group and control group. The Intervention group provided Occupational therapy based on the MOHO theory.
  Occupational therapy based on the MOHO theory: We selected two acute wards in the Songde hospital as the intervention group and the control group. At the same time, the demographic data of the participants were collected, including gender, age, age of onset, marital status, education level, work experience, etc., and the clinical records, including assessment of mental symptoms and medication records, etc. Continuity or categorical information on Occupational performance, personal and social performance, instrumental activities daily living, and clinical performance.
- Control Group: In order to indicate the occupation identity and competence to validate the OT@tcpc service model. We recruited 70 inpatients with schizophrenia and divided into intervention group and control group. The control group adopted the original Occupational therapy model.
  At the same time, the demographic data of the participants were collected, including gender, age, age of onset, marital status, education level, work experience, etc., and the clinical records, including assessment of mental symptoms and medication records, etc. Continuity or categorical information on Occupational performance, personal and social performance, instrumental activities daily living, and clinical performance.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9) | 43.4 (9.4) | 43.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Onset age [Mean (Standard Deviation); unit: years] | 20.1 (4.8) | 19.0 (3.8) | 19.56 (4.29)
Duration of illness [Mean (Standard Deviation); unit: years] | 23.0 (8.6) | 24.4 (8.6) | 23.7 (8.4)
Marital Status [Count of Participants; unit: Participants]
  Single | 15 | 14 | 29
  Married | 2 | 1 | 3
  Divorced | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Junior high school | 1 | 3 | 4
  Senior high school | 7 | 7 | 14
  College and above | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Occupational Performance History Interview-II (OPHI-II) Total and Subscale Scores
Description: The Occupational Performance History Interview-Second Version(OPHI-II) was tested before and after in the intervention group and the control group to explain the intervention effect of the MOHO theory-based treatment model.
  OPHI-II is a semi-structured interview that gathers life history information. The OPHI-II contains 3 sub-domains: OPHI-II Occupational Identity(range 11~44)、OPHI-II Occupational Competence(range 9~36)、OPHI-II Occupational Behavior Settings(range 9~36).
  The three sub-domains are divided into 4 levels, in which 4 points indicate good performance, 3 points indicate good functions, 2 points indicate lack of certain functions, and 1 points indicate poor functions. The total score of OPHI-II is equal to the sum of the three sub-domains (scores 29 to 116; higher scores indicate higher performance).
Time Frame: 2 weeks
Population: Individuals with schizophrenia were recruited from acute ward of the Psychiatric Department of Taipei City Hospital.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 17 | 16
score on a scale
  OPHI-II Total score (pretest) | 66.2 (8.0) | 69.4 (6.8)
  OPHI-II Occupational Identity (pretest) | 24.9 (4.8) | 25.7 (3.4)
  OPHI-II Occupational Competence (pretest) | 20.7 (2.6) | 22.1 (2.3)
  OPHI-II Occupational Behavior Settings (pretest) | 20.7 (2.7) | 21.6 (2.3)
  OPHI-II Total score (posttest 2 weeks) | 67.1 (8.3) | 67.6 (7.3)
  OPHI-II Occupational Identity (posttest 2 weeks) | 25.3 (5.3) | 25.0 (3.8)
  OPHI-II Occupational Competence (posttest 2 weeks) | 20.9 (2.7) | 21.5 (2.0)
  OPHI-II Occupational Behavior Settings (posttest 2 weeks) | 20.9 (2.2) | 21.1 (2.6)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Statistical Anaiysis 1 is according to Occupational Performance History Interview - II (OPHI-II) total score; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [1.65 to 5.55], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Statistical Analysis 2 is based on Occupational Identity(range 11~44；higher scores indicates better performance), a sub-domain of OPHI-II. The Occupational Identity scale is designed to measure the degree to which a client has internalized a positive occupational identity (i.e., has values, interests, and confidence; sees self in various occupational roles; has an image of the kind of life desired); Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.23 to 2.37], Standard Error of Mean 0.53
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Statistical Analysis 3 is based on Occupational Competence(range 9~36；higher scores indicate better performance), a sub-domain of OPHI-II. The Occupational Competence scale is designed to measure the degree to which a client is able to sustain a pattern of occupational behavior that is productive and satisfying; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.38 to 2.11], Standard Error of Mean 0.43
Statistical Analysis 4: Comparison: Intervention Group vs Control Group; Statistical Analysis 4 is based on Occupational Behavior Settings(range 9~36；higher scores indicate greater performance), a sub-domain of OPHI-II. The Occupational Behavior Settings scale addresses the impact of the environment on the person's occupational life; Test type: Superiority; p = 0.136, Mixed Models Analysis; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.19 to 1.35], Standard Error of Mean 0.38

2. Secondary Outcome: Occupational Therapy Evaluation Scales Measure
Description: Except for Mini-Menlal State Examination(MMSE), all other tools were tested before and after in the intervention group and the control group to explain the intervention effect of the MOHO theory-based treatment model
  The secondary outcome included the following instruments:
  1. Mini-Menlal State Examination, MMSE(range 0~30；the higher scores indicate greater ability)
  2. Canadian Occupational Performance Measure, COPM(performance and satisfaction, each range 1~10；the higher scores indicate greater performance)
  3. Personal and Social Performance scale , PSP(range 1~100；the higher scores indicate greater performance)
  4. Clinical Global Impressions Scale of Severity, CGIS(range 1~7；the lower scores indicate greater performance)
  5. Comprehensive Occupational Therapy Evaluation Scale, COTES(range 20~100；the higher scores indicate greater performance)
  6. Lawton Instrumental Activities Daily Living, LIADL(range 0~23；the higher scores indicate greater performance)
Time Frame: 2 weeks
Population: Individuals with schizophrenia were recruited from acute ward of the Psychiatric Department of Taipei City Hospital.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 17 | 16
score on a scale
  MMSE(pretest) | 27.5 (2.5) | 27.8 (2.5)
  CGIS(pretest) | 3.9 (0.8) | 4.0 (0.9)
  LIADL(pretest) | 18.1 (4.8) | 17.8 (4.2)
  COTES(pretest) | 70.8 (7.9) | 74.9 (7.8)
  COPM-C performance(pretest) | 5.7 (2.6) | 5.1 (2.3)
  COPM-C satisfaction(pretest) | 5.5 (2.9) | 4.8 (2.5)
  PSP(pretest) | 52.1 (15.9) | 51.9 (12.5)
  CGIS(posttest 2 weeks) | 3.6 (1.0) | 3.4 (1.0)
  LIADL(posttest 2 weeks) | 18.2 (4.3) | 18.6 (3.0)
  COTES(posttest 2 weeks) | 71.9 (7.1) | 74.3 (8.6)
  COPM-C performance(posttest 2 weeks) | 6.2 (2.5) | 5.1 (2.3)
  COPM-C satisfaction(posttest 2 weeks) | 6.2 (2.6) | 4.7 (2.4)
  PSP(posttest 2 weeks) | 53.4 (15.4) | 55.4 (11.3)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Statistical Analysis 1 is based on Lawton Instrumental Activities Daily Living (range 0~23；the higher scores indicate greater performance) total scores; Test type: Superiority; p = 0.592, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.90 to 2.25], Standard Error of Mean 1.53
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Statistical Analysis 2 is based on Comprehensive Occupational Therapy Evaluation Scale (range 20~100；the higher scores indicate greater performance) total scores; Test type: Superiority; p = 0.302, Mixed Models Analysis; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-2.29 to 7.23], Standard Error of Mean 2.37
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; Statistical Analysis 3 is based on Personal and Social Performance scale (range 1~100；the higher scores indicate greater performance) total scores; Test type: Superiority; p = 0.931, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-6.25 to 6.82], Standard Error of Mean 3.25
Statistical Analysis 4: Comparison: Intervention Group vs Control Group; Statistical Analysis 4 is based on Canadian Occupational Performance Measure (range 1~10；the higher scores indicate greater performance) total scores; Test type: Superiority; p = 0.981, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-1.73 to 1.69], Standard Error of Mean 0.85

ADVERSE EVENTS:
Time Frame: two weeks
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT04465422/Prot_SAP_000.pdf